CLINICAL TRIAL: NCT06813365
Title: A Phase 1, Open-Label, Multicenter Study to Assess the Safety, Tolerability, Pharmacokinetics, and Anti-tumor Efficacy of DZD6008 in Patients With Advanced Non-Small Cell Lung Cancer (NSCLC) With EGFR Mutation (TIAN-SHAN2)
Brief Title: Assessing an Oral EGFR Inhibitor, DZD6008 in Patients Who Have Advanced NSCLC With EGFR Mutations (TIAN-SHAN2)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dizal Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DZ2023C0002
Record Dates: First submitted 2024-12-23; First posted 2025-02-06 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Nonsmall-cell Lung Cancer
Keywords: Lung Cancer, EGFR mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (10):
- Part A Dose Escalation cohorts (20 mg once daily [QD]) (Experimental)
  Interventions: Drug: DZD6008
- Part A Dose Escalation cohorts (40 mg QD) (Experimental)
  Interventions: Drug: DZD6008
- Part A Dose Escalation cohorts (60 mg QD) (Experimental)
  Interventions: Drug: DZD6008
- Part A Dose Escalation cohorts (90 mg QD) (Experimental)
  Interventions: Drug: DZD6008
- Part A Dose Escalation cohorts (120 mg QD) (Experimental)
  Interventions: Drug: DZD6008
- Part A Dose Escalation cohorts (150 mg QD) (Experimental)
  Interventions: Drug: DZD6008
- Part B Dose Expansion cohorts (selected dose 1 QD) (Experimental)
  Interventions: Drug: DZD6008
- Part B Dose Expansion cohorts (selected dose 2 QD) (Experimental)
  Interventions: Drug: DZD6008
- Food effect cohort (selected dose 1) (Experimental)
  Interventions: Drug: DZD6008
- Food effect cohort (selected dose 2) (Experimental)
  Interventions: Drug: DZD6008

INTERVENTIONS:
Drug: DZD6008 — Daily dose of DZD6008

SUMMARY:
This study is designed to evaluate safety and antitumor activity of DZD6008 in patients with advanced NSCLC with EGFR mutations. This is the first time the drug is tested in human.

DETAILED DESCRIPTION:
The study includes two parts: Part A (dose escalation) and Part B (dose expansion). In Part A, locally advanced or metastatic NSCLC patients with EGFR sensitizing mutations (Exon19del and/or L858R) following at least 1 prior EGFR TKI and platinum-based chemotherapy will be enrolled. In Part B, locally advanced or metastatic NSCLC patients with EGFR sensitizing mutations following 1 prior third-generation EGFR TKI and who are treatment naïve will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be able to provide documented informed consent.
2. Aged ≥ 18 years.
3. Histologically or cytologically confirmed diagnosis of NSCLC, locally advanced or metastatic, not suitable for curative therapy.
4. Documentation of EGFR sensitizing mutation (Exon19del and/or L858R) from a local CLIA-certified laboratory (or equivalent).
5. Provide adequate amount of pretreatment tumor samples for retrospective confirmation of EGFR mutations by the central laboratory.
6. Part A: Failed (progressed or are intolerant) at least 1 prior EGFR TKI and platinum-based chemotherapy. Part B: Cohorts 1 and 2: Failed 1 prior third-generation EGFR TKI. Cohorts 3 and 4: Patients who are treatment naïve.

   Note: Patients enrolled in the study should be representative of the population to meet the need for efficacy analysis in the population after TKI failure (e.g., including appropriate proportion and number of patients with the C797X mutation if possible)
7. ECOG 0 or 1 with predicted life expectancy ≥ 12 weeks.
8. Patients with brain metastases must have a stable BM status.
9. Measurable disease per RECIST 1.1.
10. Adequate hematopoietic and other organ system functions.
11. Male Patients with female partners of childbearing potential should use barrier contraceptives and refrain from donating sperm during their participation in this study and for 3 months following the last dose of the study drug.

Exclusion Criteria:

1. Carry any other known EGFR alterations, including but not limited to uncommon EGFR mutations (G719X, S768I, L861Q, exon 20 insertions, etc.)(Part B).
2. NSCLC with mixed small cell lung cancer (SCLC) or NSCLC with histologic SCLC transformation.
3. Prior treatment with any of the following:1)Immunotherapy or other antibody therapy within 4 weeks prior to the first administration;2)Any cytotoxic chemotherapy, investigational drugs or other anticancer drugs from a previous treatment regimen or clinical study within 14 days prior to the first administration;3)Radiotherapy with a limited field of radiation for palliation within 7 days of the first dose, radiation to more than 30% of the bone marrow or with a wide field of radiation within 28 days before screening;4)Currently receiving or unable to stop drug or herbal supplements known to be potent inhibitors or inducers of cytochrome P450 (CYP)3A4. A washout period of at least 2 weeks for strong inhibitors and 3 weeks for strong inducers is required prior to the first study drug administration.5)currently receiving or unable to stop drugs known to be CYP3A4 sensitive substrate with a narrow therapeutic index. A washout period of at least 14 days is required prior to the first study drug administration;6)currently receiving or unable to stop drugs known to be proton pump inhibitors. A washout period of at least 7 days is required prior to the first study drug administration;7)Major surgery within 4 weeks of the first administration of DZD6008 or anticipated during the study period.
4. Any unresolved toxicities from prior anti-cancer therapy greater than CTCAE Grade 1.
5. Spinal cord compression or leptomeningeal metastasis.
6. Patients with any other malignancy within 2 years of the first administration of study drug.
7. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses as judged by investigator.
8. Patients with active infection including but not limited to HBV, HCV, HIV and active infection of COVID-19.
9. Resting QTcF > 470 msec; Any clinically significant abnormalities in rhythm, conduction or morphology of resting ECG;Any factors that increase the risk of QTc prolongation.
10. Past medical history of ILD or active ILD.
11. Diseases which would preclude adequate absorption of DZD6008.
12. Women who are pregnant or breastfeeding.
13. Hypersensitivity to active or inactive excipients of DZD6008.
14. Involvement in the planning and conduct of the study.
15. Judgment by the investigator that the patients is unlikely to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Part A: To assess safety and tolerability | 21 days after the first multiple dose.
  Number of participants with Dose-limiting Toxicities (DLTs)
Part A: To assess safety and tolerability | Through the study completion, an average of around 1 year.
  Number of participants with Adverse events (AEs)/Serious adverse events (SAEs)
Part B: To assess anti-tumor activity | Through the study completion, an average of around 1 year.
  Objective Response Rate (ORR) as assessed by investigators per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

SECONDARY OUTCOMES:
Part A: To characterize the plasma concentration of DZD6008 following single and multiple oral dose administration | From first dosing to cycle 7 day 1, each cycle is 21 days.
  Total concentrations of DZD6008 in plasma.
Part A: To assess the urine concentration of DZD6008 | At the first day of cycle 2 (each cycle is 21 days).
  Total concentrations of DZD6008 in urine.
Part A: To assess cerebrospinal fluid of DZD6008 in participants with brain metastasis at baseline | Cycle 1 day 15.
  Total concentrations of DZD6008 in cerebrospinal fluid
Part A: To assess the effect of low-fat food on the plasma concentration of DZD6008 | The first dosing day on cycle 0 (cycle 0 is 3 days).
  Total concentrations of DZD6008 in plasma.
Part A: To assess the anti-tumor activity | Through the study completion, an average of around 1 year.
  ORR as assessed by investigators per RECIST version 1.1.
Part A: To assess the anti-tumor activity | Through the study completion, an average of around 1 year.
  Duration of Response (DoR) as assessed by investigators per RECIST version 1.1.
Part A: To assess the anti-tumor activity | Through the study completion, an average of around 1 year.
  Progression Free Survival (PFS) as assessed by investigators per RECIST version 1.1.
Part B: To assess the anti-tumor activity | Through the study completion, an average of around 1 year.
  Progression ORR as assessed by Independent Review Committee (IRC) per RECIST version 1.1.
Part B: To assess the anti-tumor activity | Through the study completion, an average of around 1 year.
  Progression DoR as assessed by IRC and investigators per RECIST version 1.1.
Part B: To assess the preliminary anti-tumor activity | Through the study completion, an average of around 1 year.
  Progression PFS as assessed by IRC and investigators per RECIST version 1.1.
Part B: Plasma concentration of DZD6008 | From first dosing to cycle 11 day 1, each cycle is 21 days.
  Total concentrations of DZD6008 in plasma.
Part B: To assess safety and tolerability | Through the study completion, an average of around 1 year.
  Number of participants with Adverse events (AEs)/Serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided